CLINICAL TRIAL: NCT05607771
Title: Paired Non-inferiority Study Comparing Overture Semi-Automated Vitrification System ("DaVitri") to Standard Manual Process
Brief Title: DaVitri: Semi-Automated Vitrificacion Clinical Study
Acronym: DaVitri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Overture Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: CIP-DV-000-GEN-001
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Fertility Issues
Keywords: Vitrification
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual (Experimental): Oocytes will be prepared for vitrification using the manual protocol
  Interventions: Device: Manual Vitrification
- Automated (Experimental): Oocytes will be prepared for vitrification using Davitri device
  Interventions: Device: Automated Vitrification

INTERVENTIONS:
Device: Manual Vitrification — Oocytes will be prepared for vitrification using the manual protocol
  Arms: Manual
Device: Automated Vitrification — Oocytes will be prepared for vitrification using the DaVitri device
  Arms: Automated

SUMMARY:
The main objective of this clinical study is to demonstrate the non-inferiority of the semi automated device (DaVitri) developed by Overture Life in the preparation procedures for vitrification of human samples.

DETAILED DESCRIPTION:
Vitrification is a manual technique that is routinely used in assisted reproduction clinics for the cryopreservation of oocytes and embryos in liquid nitrogen at -196oC. There are different methods of vitrification, the most used being the Cryotop of Kitazato. This is a manual process that requires precision and experience to achieve a good result. For this reason, the correct execution of the technique is considered key in in vitro fertilization (IVF) treatments, as it can favor the preservation of fertility and optimize clinical results.

The purpose of the study is to validate the viability of the semi automated vitrification process, to obtain survival rates similar to or superior to manual processes, and also the capacity to provide greater reproducibility in the results.

The semi automatic exchange of vitrification fluids in human oocytes is as efficient as the manual procedure, in terms of survival (85-90%), but with significantly lower variability between technicians and between centers (95% reproducibility), as well as reduced manual processing times.

The initial hypothesis is that semi automated vitrification equals or improves the manual technique, thus introducing a new standardized protocol for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Donors will be selected according to the clinic's usual inclusion criteria in terms of infectious diseases, genetic diseases, karyotype, etc.

Exclusion Criteria:

* BMI<18.5 or BMI >25
* Implantation failure
* Abnormal ovulation cycle
* Endometrial thickness > 7mm

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Thaw survival rates of oocytes | Day 1
  Number of valid oocytes/numbers of randomized oocytes

SECONDARY OUTCOMES:
Blastocyst formation rate | Day 5
  Number of blastocysts at day 5 or 6/number of fertilized oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Neuspiller, MD, Principal Investigator — WeFiv
Locations (2):
- Argentina (2):
  - WeFIV Buenos Aires, Buenos Aires
  - Halitus Instituto Médico, Buenos Aires

IPD SHARING:
Plan to Share IPD: No